CLINICAL TRIAL: NCT04814888
Title: Prediction of Endotracheal Tube Size Using a Printed Three-dimensional Airway Model in Pediatric Patients With Congenital Heart Disease: a Prospective, Single-center, Single- Group Study
Brief Title: 3D Airway Model for Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Clinical associate professor, Pusan National University Yangsan Hospital
Other Study IDs: 05-2019-116
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: intubation with a cuffed ETT by a printed 3D airway model — Two anaesthesiologists unaware of patient's demographic data such as patient's height, weight, and age predicted and recorded ETT size by inserting various sized cuffed-ETTs (MallinckrodtTM Hi-Lo tracheal tube, Covidien, Ireland) to a printed 3D airway model. If the diameter of trachea undersized, air leak around ETT can occur. In that case, we can use that ETT after inflating the pilot balloon with small amount of air. Standard monitoring (non-invasive blood pressure measurement, electrocardiogram, and pulse oximetry) was applied to pediatric patients in the operating room and general anesthesia was induced with ketamine 1 mg/kg and rocuronium 0.6 mg/kg and maintained with sevoflurane. After intubation with a cuffed ETT by a printed 3D airway model was finished, an air leak test was performed by one of three anaesthesiologists dedicated to pediatric cardiac anesthesia.

SUMMARY:
To determine the correct size of endotracheal tubes (ETT) for endotracheal intubation of pediatric patients is no menial task. Although new methods have been investigated to determine ETT size, and the three-dimensional (3D) printing technology has been successful in the field of surgery, there are not many studies in the field of anesthesia. The purpose of this study is to evaluate the accuracy of a 3D airway model for prediction of the correct ETT size, and compare the results with a conventional age-based formula in pediatric patients.

DETAILED DESCRIPTION:
To determine the correct size of endotracheal tubes (ETT) for endotracheal intubation of pediatric patients is no menial task. Although new methods have been investigated to determine ETT size, and the three-dimensional (3D) printing technology has been successful in the field of surgery, there are not many studies in the field of anesthesia. The purpose of this study is to evaluate the accuracy of a 3D airway model for prediction of the correct ETT size, and compare the results with a conventional age-based formula in pediatric patients. : Thirty five pediatric patients under 6 years of age who were scheduled for congenital heart surgery. In the pre-anaesthetic period, the patient's computed tomography (CT) images were converted to STL files using the 3D conversion program. An FDM type 3D printer was used to print 3D airway models from the sub-glottis to the upper carina. ETT size was selected by inserting various sized cuffed-ETTs to a printed 3D airway model.

ELIGIBILITY:
Inclusion Criteria:

* children under 6 years of age (range 4 days to 61 months) scheduled for surgery for congenital heart disease with chest computed tomography (CT) images including upper airways

Exclusion Criteria:

* pediatric patients with intubation or tracheostomy before general anesthesia due to underlying disease
* small sized airway with inner diameter <3.0 mm because of pre-term or low birth weight
* unstable vital signs during induction
* history of difficult intubation
* emergency surgery where printing a 3D airway model in advance was not possible

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We enrolled children under 6 years of age (range 4 days to 61 months) scheduled for surgery for congenital heart disease with chest computed tomography (CT) images including upper airways from September 3, 2019, to March, 16, 2020. Pediatric patients with congenital heart disease were chosen because they usually keep their ETT with mechanical ventilation in the intensive care unit and also have relatively high risk of complication associated with ETT comparing to healthy patients. Therefore, we think it is more important to select appropriate size of ETT in pediatric patients with congenital heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
ETT size prediction by the printed 3D airway model | during anesthesia induction
  The reliability of ETT size prediction by the printed 3D airway model was compared with the results of the age-based formula.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, Principal Investigator — Department of Anesthesia and Pain Medicine, School of Medicine, Pusan National University
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No